CLINICAL TRIAL: NCT01885585
Title: Eliquis (Apixaban) Regulatory Post Marketing Surveillance in Clinical Practice for Venous Thromboembolism (VTE) Prevention
Brief Title: Eliquis Regulatory Post Marketing Surveillance (rPMS)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-222
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with risk of VTE: Patients undergoing elective total hip replacement arthroplasty or elective total knee replacement arthroplasty and signed on the data release
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: Eliquis

SUMMARY:
The objective of this regulatory Post-Marketing Surveillance in Korea is to reconfirm the clinical usefulness of Eliquis through collecting, reviewing, identifying and verifying the safety and effectiveness information about Eliquis in general practice

ELIGIBILITY:
Inclusion Criteria:

* Signed data release
* Patients undergoing elective total hip replacement arthroplasty or elective total knee replacement arthroplasty

Exclusion Criteria:

* Being treated for an indication not approved for the use of Eliquis® in Korea
* Is contraindicated for the use of Eliquis® as described in the Korean label

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic Patients must be ≥19 years of age, at risk for venous thrombosis, and have elected to undergo total hip replacement arthroplasty or total knee replacement arthroplasty will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) and serious AEs | Up to 30 days after last study drug dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Seoul, South Korea

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx